CLINICAL TRIAL: NCT00558896
Title: A Phase II Trial of CC-4047 Plus Dexamethasone in Patients With Relapsed of Refractory Multiple Myeloma or Amyloidosis
Brief Title: CC-4047 and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma or Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574742; P30CA015083 (NIH); 07-003064 (Other: Mayo Clinic IRB); NCI-2009-01283 (Registry Identifier: NCI-CTRP); MC0789 (Other: Mayo Clinic Cancer Center); NCT01219634 (obsolete NCT alias)
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Relapsed Myeloma (<4 Prior Regimens) (Experimental): Pomalidomide: 2 mg orally once daily, days 1-28 of 28 day cycle
  Dexamethasone: 40 mg on days 1, 8, 15 ad 22 of 28 day cycle
  Interventions: Drug: dexamethasone; Drug: pomalidomide
- Lenalidomide Refractory Myeloma (Experimental): Pomalidomide: 2 mg orally once daily, days 1-28 of 28 day cycle
  Dexamethasone: 40 mg on days 1, 8, 15 ad 22 of 28 day cycle
  Interventions: Drug: dexamethasone; Drug: pomalidomide
- Bortezomib/Lenalidomide Refractory/Relapsed Myeloma (Experimental): Pomalidomide: 2 mg orally once daily, days 1-28 of 28 day cycle
  Dexamethasone: 40 mg on days 1, 8, 15 ad 22 of 28 day cycle
  Interventions: Drug: dexamethasone; Drug: pomalidomide
- Bortezomib/Lenalidomide Relapsed/Refractory Myeloma (Experimental): Pomalidomide: 4 mg orally once daily, days 1-28 of 28 day cycle
  Dexamethasone: 40 mg on days 1, 8, 15 ad 22 of 28 day cycle
  Interventions: Drug: dexamethasone; Drug: pomalidomide
- Relapsed Myeloma (< 4 Prior Regimens) (Experimental): Pomalidomide: 4 mg orally once daily, days 1-28 of 28 day cycle
  Dexamethasone: 40 mg on days 1, 8, 15 ad 22 of 28 day cycle
  Interventions: Drug: dexamethasone; Drug: pomalidomide
- Relapsed/Refractory Myeloma (Experimental): Pomalidomide: 4 mg orally once daily, days 1-21 of 28 day cycle
  Dexamethasone: 40 mg on days 1, 8, 15 ad 22 of 28 day cycle
  Interventions: Drug: dexamethasone; Drug: pomalidomide
- Relapsed Amyloidosis (Experimental): Pomalidomide: 2 mg orally once daily, days 1-28 of 28 day cycle
  Dexamethasone: 40 mg on days 1, 8, 15 ad 22 of 28 day cycle
  Interventions: Drug: dexamethasone; Drug: pomalidomide

INTERVENTIONS:
Drug: dexamethasone — 40 mg/day administered through PO (with food) at Days 1, 8, 15, 22 per cycle.
Drug: pomalidomide — 2 or 4 mg/day administered through PO at days 1 - 28 or days 1-21 (see Arm description for specific dosing).
  Other Names: CC-4047

SUMMARY:
RATIONALE: Biological therapies, such as CC-4047, may stimulate the immune system in different ways and stop cancer cells from growing. Dexamethasone and CC-4047 may stop the growth of cancer cells by blocking blood flow to the cancer. Giving CC-4047 together with dexamethasone may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving CC-4047 together with dexamethasone works in treating patients with relapsed or refractory multiple myeloma or amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the response rate and duration of remission with low-dose CC-4047 plus dexamethasone in patients with relapsed or refractory multiple myeloma or amyloidosis.
* To assess the toxicity of CC-4047 plus dexamethasone in this patient population.
* To assess in an expansion cohort the response rate with an increase in CC-4047 dose among patients who fail to respond adequately to the initial starting dose following the first 2 courses of treatment.
* To assess the response rate and duration of remission with CC-4047 plus dexamethasone in patients with lenalidomide resistant or refractory multiple myeloma.
* To assess the response rate and duration of remission with CC-4047 plus dexamethasone in patients with previously treated light chain amyloidosis.
* To assess the response rate and duration of remission with low- and high-dose CC-4047 plus dexamethasone in patients with lenalidomide and bortezomib refractory multiple myeloma.
* To assess the response rate and duration of remission with high-dose CC-4047 plus dexamethasone in patients with relapsed or refractory myeloma who received ≤ 3 treatment regimens.

OUTLINE: Patients are grouped according to disease status (relapsed/refractory myeloma [closed to accrual as of 8/5/2008] vs lenalidomide resistant/refractory myeloma [closed to accrual as of 4/2/2009] vs previously treated light chain amyloidosis vs lenalidomide and bortezomib resistant/refractory myeloma {low-dose/day}[closed to accrual as of 11/20/09] vs lenalidomide and bortezomib resistant/refractory myeloma (high-dose/day) vs relapsed/refractory myeloma {high-dose/day}).

Patients receive oral CC-4047 on days 1-28 and oral dexamethasone on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 4 weeks and then at 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Symptomatic multiple myeloma
* Previously treated disease meeting one of the following criteria:

  * Have light-chain amyloidosis that has been treated with at least one prior regimen
  * Symptomatic (relapsed or refractory) multiple myeloma

    * Patients must have received 1-3 treatment regimens
    * Induction therapy followed by autologous stem cell transplantation and consolidation considered one regimen
* Measurable disease, as defined by 1 of the following:

  * Serum monoclonal protein ≥ 1.0 g by protein electrophoresis
  * More than 200 mg of monoclonal protein in the urine on 24-hour electrophoresis
  * Serum immunoglobulin free light chain (FLC) > 10 mg/dL and an abnormal FLC ratio
  * Measurable soft tissue plasmacytoma, not previously irradiated
  * More than 30% plasma cells in bone marrow
* At least 10% plasma cells as measured by bone marrow aspirate, bone marrow biopsy, or labeling index
* No monoclonal gammopathy of undetermined significance (not applicable for patients with amyloid)
* No smoldering myeloma (not applicable for patients with amyloid)

PATIENT CHARACTERISTICS:

* ECOG performance status 0, 1, or 2
* ANC ≥ 1,000/μL
* Platelet count ≥ 75,000/μL
* Creatinine ≤ 2.5 mg/dL
* Not pregnant or nursing

  * Women must refrain from breastfeeding during study participation and for at least 28 days after discontinuation of study drug
* Negative pregnancy test
* Fertile female patients must use two reliable forms of contraception simultaneously at least 28 days before beginning, during, and at least 28 days after completion of study drug

  * The two methods of reliable contraception must include one highly effective method (i.e., intrauterine device [IUD], hormonal [birth control pills, injections, or implants], tubal ligation, or partner's vasectomy) and one additional effective (barrier) method (i.e., latex condom, diaphragm, or cervical cap)
* Fertile male patients must use a latex condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 28 days after stopping treatment
* Men must agree to abstain from donating semen or sperm during study participation and for 28 days after discontinuation of study drug
* Willing to abstain from donating blood during study participation and for 28 days after discontinuation of study drug
* No uncontrolled infection
* No other active malignancy
* No New York Heart Association class III or IV cardiac disease (all patients)

  * Serum troponin T > 0.10 ng/mL (amyloid patients only)
* No known positivity for HIV or active hepatitis infection
* No active deep vein thrombosis or pulmonary embolism that has not been therapeutically anticoagulated
* No condition, including the presence of laboratory abnormalities, that places the patient at unacceptable risk for participating in the study or confounds the ability to interpret data from the study
* No known hypersensitivity to thalidomide or lenalidomide including development of erythema nodosum if characterized by a desquamating rash
* No peripheral neuropathy > grade 2

PRIOR CONCURRENT THERAPY:

* All previous cancer therapy, including chemotherapy and investigational agents, must have been discontinued ≥ 2 weeks prior to study registration
* No radiotherapy ≤ 14 days prior to study registration
* No other concurrent anti-myeloma therapy
* No concurrent radiotherapy, except for palliation of a single painful bone lesion or fracture
* Routine concurrent bisphosphonate therapy allowed for patients with myeloma bone disease
* Willing and able to take aspirin or alternate prophylactic anticoagulation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Q. Lacy, MD, Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Dispenzieri A, Buadi F, Laumann K, LaPlant B, Hayman SR, Kumar SK, Dingli D, Zeldenrust SR, Mikhael JR, Hall R, Rajkumar SV, Reeder C, Fonseca R, Bergsagel PL, Stewart AK, Roy V, Witzig TE, Lust JA, Russell SJ, Gertz MA, Lacy MQ. Activity of pomalidomide in patients with immunoglobulin light-chain amyloidosis. Blood. 2012 Jun 7;119(23):5397-404. doi: 10.1182/blood-2012-02-413161. Epub 2012 Apr 4. PMID 22493299
- [Derived] Lacy MQ, Allred JB, Gertz MA, Hayman SR, Short KD, Buadi F, Dispenzieri A, Kumar S, Greipp PR, Lust JA, Russell SJ, Dingli D, Zeldenrust S, Fonseca R, Bergsagel PL, Roy V, Stewart AK, Laumann K, Mandrekar SJ, Reeder C, Rajkumar SV, Mikhael JR. Pomalidomide plus low-dose dexamethasone in myeloma refractory to both bortezomib and lenalidomide: comparison of 2 dosing strategies in dual-refractory disease. Blood. 2011 Sep 15;118(11):2970-5. doi: 10.1182/blood-2011-04-348896. Epub 2011 Jun 20. PMID 21690557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2007 and March 2012, 7 sequential phase 2 trials (reported as separate arms) were conducted. A total of 378 participants were recruited at Mayo Clinic (Arizona, Florida or Arizona).
Pre-assignment Details: One patient was deemed ineligible and excluded from all analyses.
Groups:
- Relapsed Myeloma (<4 Prior Regimens): Low Dose; Lenalidomide Refractory Myeloma: Low Dose; Bortezomib/Lenalidomide Refractory/Relapsed Myeloma: Low Dose; Relapsed Amyloidosis: Low Dose: Pomalidomide: 2 mg orally once daily, days 1-28 of 28 day cycle
  Dexamethasone: 40 mg on days 1, 8, 15 ad 22 of 28 day cycle
- Bortezomib/Lenalidomide Relapsed/Refractory Myeloma: High Dose; Relapsed Myeloma (< 4 Prior Regimens): High Dose: Pomalidomide: 4 mg orally once daily, days 1-28 of 28 day cycle
  Dexamethasone: 40 mg on days 1, 8, 15 ad 22 of 28 day cycle
- Relapsed/Refractory Myeloma: High Dose: Pomalidomide: 4 mg orally once daily, days 1-21 of 28 day cycle
  Dexamethasone: 40 mg on days 1, 8, 15 ad 22 of 28 day cycle
Period: Overall Study
Arm/Group | Relapsed Myeloma (<4 Prior Regimens): Low Dose | Lenalidomide Refractory Myeloma: Low Dose | Bortezomib/Lenalidomide Refractory/Relapsed Myeloma: Low Dose | Bortezomib/Lenalidomide Relapsed/Refractory Myeloma: High Dose | Relapsed Myeloma (< 4 Prior Regimens): High Dose | Relapsed/Refractory Myeloma: High Dose | Relapsed Amyloidosis: Low Dose
Started | 60 | 34 | 35 | 35 | 60 | 120 | 33
Completed | 39 | 27 | 30 | 23 | 37 | 68 | 9
Not Completed | 21 | 7 | 5 | 12 | 23 | 52 | 24
Not completed — Adverse Event | 1 | 1 | 1 | 3 | 4 | 10 | 3
Not completed — Death | 3 | 0 | 2 | 3 | 2 | 2 | 6
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1 | 1 | 5 | 5
Not completed — Alternative Treatment | 2 | 2 | 0 | 2 | 6 | 7 | 1
Not completed — Physician discretion | 3 | 2 | 1 | 2 | 1 | 3 | 3
Not completed — Continues on treatment | 10 | 1 | 0 | 1 | 9 | 25 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relapsed Myeloma (<4 Prior Regimens): Low Dose | Lenalidomide Refractory Myeloma: Low Dose | Bortezomib/Lenalidomide Refractory/Relapsed Myeloma: Low Dose | Bortezomib/Lenalidomide Relapsed/Refractory Myeloma: High Dose | Relapsed Myeloma (< 4 Prior Regimens): High Dose | Relapsed/Refractory Myeloma: High Dose | Relapsed Amyloidosis: Low Dose | Total
Number analyzed (Participants) | 60 | 34 | 35 | 35 | 60 | 120 | 33 | 377
Age, Continuous [Median (Full Range); unit: years] | 65.5 [35 to 88] | 61.5 [39 to 77] | 62 [39 to 77] | 61 [45 to 77] | 65.5 [32 to 82] | 65 [36 to 85] | 66 [52 to 82] | 64 [32 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 11 | 8 | 14 | 20 | 47 | 14 | 138
  Male | 36 | 23 | 27 | 21 | 40 | 73 | 19 | 239
Region of Enrollment [Number; unit: participants]
  United States | 60 | 34 | 35 | 35 | 60 | 120 | 33 | 377

OUTCOME MEASURES:

1. Primary Outcome: The Number of Confirmed Hematologic Responses (Complete, Partial, or Very Good Partial Response)
Description: Response that was confirmed on 2 consecutive evaluations
  * Complete Response(CR): Complete disappearance of M-protein from serum and urine on immunofixation, normalization of Free Light Chain (FLC) ratio and <5% plasma cells in bone marrow.
  * Very Good Partial Response(VGPR): >=90% reduction in serum M-component; Urine M-Component <100mg per 24hours; <=5% plasma cells in bone marrow.
  * Partial Response(PR): >=50% reduction in serum M-component and/or Urine M-Component >=90% reduction or <200mg per 24hours; or >=50% decrease in difference between involved and uninvolved FLC levels.
Time Frame: Duration of study (up to 3 years)
Measure: Number; unit: participants
Arm/Group | Relapsed Myeloma (<4 Prior Regimens): Low Dose | Lenalidomide Refractory Myeloma: Low Dose | Bortezomib/Lenalidomide Refractory/Relapsed Myeloma: Low Dose | Bortezomib/Lenalidomide Relapsed/Refractory Myeloma: High Dose | Relapsed Myeloma (< 4 Prior Regimens): High Dose | Relapsed/Refractory Myeloma: High Dose | Relapsed Amyloidosis: Low Dose
Number analyzed (Participants) | 60 | 34 | 35 | 35 | 60 | 120 | 33
participants | 39 | 11 | 9 | 10 | 23 | 25 | 16

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from registration to progression or death due to any cause. PFS was analyzed using Kaplan Meier method.
  Progression was defined as any one or more of the following:
  * 25% increase in serum M-component (absolute increase >= 0.5g/dl)
  * 25% increase in urine M-component (absolute increase >= 200mg/24hour
  * 25% increase in the difference between involved and uninvolved Free Light Chain levels (absolute increase >= 10mg/dl)
  * 25% increase in bone marrow plasma cell percentage (absolute increase of >=10%)
  * Definite development of new bone lesion or soft tissue plasmacytomas
Time Frame: Duration of study (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Relapsed Myeloma (<4 Prior Regimens): Low Dose | Lenalidomide Refractory Myeloma: Low Dose | Bortezomib/Lenalidomide Refractory/Relapsed Myeloma: Low Dose | Bortezomib/Lenalidomide Relapsed/Refractory Myeloma: High Dose | Relapsed Myeloma (< 4 Prior Regimens): High Dose | Relapsed/Refractory Myeloma: High Dose | Relapsed Amyloidosis: Low Dose
Number analyzed (Participants) | 60 | 34 | 35 | 35 | 60 | 120 | 33
months | 13 [8.1 to 20.4] | 5 [2.7 to 10.3] | 6.4 [3.2 to 8.0] | 3.3 [1.9 to 6.2] | 7.7 [4.8 to 10.8] | 4.3 [2.9 to 5] | 14.1 [9.7 to 21.1]

3. Secondary Outcome: Duration of Response
Description: Duration of response was calculated from the documentation (date) of first response (CR, VGPR, or PR) until the date of progression or last follow-up in the subset of patients who responded. Kaplan Meier method was used to compute this outcome.
Time Frame: Duration of study (up to 5 years)
Population: Participants who achieved a partial response(PR) or better were evaluable for this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Relapsed Myeloma (<4 Prior Regimens): Low Dose | Lenalidomide Refractory Myeloma: Low Dose | Bortezomib/Lenalidomide Refractory/Relapsed Myeloma: Low Dose | Bortezomib/Lenalidomide Relapsed/Refractory Myeloma: High Dose | Relapsed Myeloma (< 4 Prior Regimens): High Dose | Relapsed/Refractory Myeloma: High Dose | Relapsed Amyloidosis: Low Dose
Number analyzed (Participants) | 39 | 11 | 9 | 10 | 23 | 25 | 16
months | 21.3 [11.2 to 34.1] | 8.2 [3.2 to 38.4] | 15.6 [4.3 to 31.1] | 3.1 [1.8 to 14.5] | NA [NA to NA] — Median duration of response was not attained | 8.3 [4.5 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment | 19 [8.3 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment

ADVERSE EVENTS:
Description: One participant in the Relapse/Refractory Myeloma: High Dose group refused prior to starting treatment, thus was not included in the adverse event analysis.
Arm/Group | Relapsed Myeloma (<4 Prior Regimens): Low Dose | Lenalidomide Refractory Myeloma: Low Dose | Bortezomib/Lenalidomide Refractory/Relapsed Myeloma: Low Dose | Bortezomib/Lenalidomide Relapsed/Refractory Myeloma: High Dose | Relapsed Myeloma (< 4 Prior Regimens): High Dose | Relapsed/Refractory Myeloma: High Dose | Relapsed Amyloidosis: Low Dose
Serious Adverse Events (participants affected / at risk) | 22/60 | 11/34 | 15/35 | 11/35 | 21/60 | 32/119 | 18/33
Other Adverse Events (participants affected / at risk) | 60/60 | 34/34 | 34/35 | 35/35 | 60/60 | 119/119 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed Myeloma (<4 Prior Regimens): Low Dose (N=60) | Lenalidomide Refractory Myeloma: Low Dose (N=34) | Bortezomib/Lenalidomide Refractory/Relapsed Myeloma: Low Dose (N=35) | Bortezomib/Lenalidomide Relapsed/Refractory Myeloma: High Dose (N=35) | Relapsed Myeloma (< 4 Prior Regimens): High Dose (N=60) | Relapsed/Refractory Myeloma: High Dose (N=119) | Relapsed Amyloidosis: Low Dose (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 2 (2) | 5 (5) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cecum perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (10) | 6 (7) | 8 (9) | 1 (2) | 7 (7) | 13 (13) | 6 (9)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intraoperative musculoskeletal injury - Joint (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 4 (4) | 5 (5) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 4 (5) | 6 (6) | 5 (5) | 2 (2)
Platelet count decreased (Investigations) | 3 (4) | 0 (0) | 2 (3) | 3 (3) | 4 (4) | 6 (6) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed Myeloma (<4 Prior Regimens): Low Dose (N=60) | Lenalidomide Refractory Myeloma: Low Dose (N=34) | Bortezomib/Lenalidomide Refractory/Relapsed Myeloma: Low Dose (N=35) | Bortezomib/Lenalidomide Relapsed/Refractory Myeloma: High Dose (N=35) | Relapsed Myeloma (< 4 Prior Regimens): High Dose (N=60) | Relapsed/Refractory Myeloma: High Dose (N=119) | Relapsed Amyloidosis: Low Dose (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 57 (707) | 34 (241) | 34 (239) | 34 (134) | 55 (348) | 115 (418) | 31 (277)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0) | 3 (7) | 0 (0) | 2 (11) | 2 (2) | 3 (5)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (6)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (20) | 1 (1) | 1 (1) | 0 (0) | 4 (12) | 3 (3) | 3 (6)
Diarrhea (Gastrointestinal disorders) | 26 (71) | 11 (57) | 11 (47) | 8 (18) | 23 (73) | 30 (49) | 16 (44)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 3 (8) | 1 (1) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 19 (38) | 10 (37) | 11 (46) | 7 (10) | 13 (37) | 31 (43) | 13 (32)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (16) | 6 (8) | 7 (28) | 4 (4) | 6 (7) | 7 (8) | 5 (7)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 9 (19) | 4 (9) | 1 (9) | 1 (1) | 4 (14) | 1 (3) | 7 (12)
Fatigue (General disorders) | 56 (718) | 32 (278) | 31 (247) | 32 (127) | 56 (440) | 111 (372) | 32 (331)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Pain (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Infection (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (8) | 3 (3) | 4 (6) | 2 (2) | 6 (6) | 7 (8) | 3 (4)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 6 (7) | 5 (6) | 1 (1) | 0 (0) | 3 (6) | 2 (2) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraoperative ocular injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (4) | 1 (1) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (3)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Leukocyte count decreased (Investigations) | 44 (243) | 27 (92) | 29 (147) | 31 (122) | 54 (266) | 103 (303) | 22 (96)
Lymphocyte count decreased (Investigations) | 6 (69) | 4 (10) | 12 (48) | 14 (41) | 32 (130) | 8 (22) | 3 (11)
Neutrophil count decreased (Investigations) | 48 (419) | 26 (113) | 29 (132) | 30 (106) | 51 (304) | 98 (284) | 21 (90)
Platelet count decreased (Investigations) | 31 (186) | 18 (87) | 30 (137) | 30 (74) | 43 (152) | 98 (262) | 19 (93)
Weight gain (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 20 (44) | 16 (23) | 10 (22) | 12 (15) | 18 (50) | 46 (70) | 12 (37)
Blood glucose increased (Metabolism and nutrition disorders) | 14 (29) | 5 (19) | 4 (12) | 2 (2) | 16 (58) | 10 (14) | 1 (1)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3) | 1 (1) | 3 (4) | 0 (0) | 3 (5) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (3) | 1 (4) | 0 (0) | 2 (2) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (4) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 3 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (7) | 3 (4) | 1 (3) | 0 (0) | 0 (0) | 2 (7) | 2 (4)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 3 (6) | 1 (3) | 1 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (9) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (5) | 0 (0) | 2 (2) | 0 (0) | 5 (6) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myelitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neurological disorder NOS (Nervous system disorders) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 45 (664) | 23 (221) | 28 (233) | 31 (120) | 42 (349) | 94 (332) | 29 (259)
Syncope (Nervous system disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 10 (12) | 2 (2) | 4 (7) | 0 (0) | 2 (6) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (9) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 4 (5) | 1 (3)
Confusion (Psychiatric disorders) | 7 (10) | 3 (7) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 6 (8) | 0 (0) | 1 (1) | 3 (7) | 2 (2) | 2 (2) | 1 (1)
Euphoria (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 11 (17) | 0 (0) | 4 (12) | 1 (1) | 9 (18) | 4 (6) | 3 (3)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bladder stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 3 (3) | 1 (1) | 5 (11) | 4 (6) | 7 (14)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrophy skin (Skin and subcutaneous tissue disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 5 (12) | 1 (4) | 0 (0) | 2 (2) | 1 (17) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (2) | 3 (3) | 3 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes